CLINICAL TRIAL: NCT03871803
Title: Betablockers Withdrawal in Patients With Heart Failure With Preserved Ejection Fraction and Chronotropic Incompetence: Effect on Functional Capacity Rationale and Study Design of a Prospective, Randomized, Controlled Trial
Brief Title: β-blockers Withdrawal in Patients With HFpEF and Chronotropic Incompetence: Effect on Functional Capacity (Preserve-HR)
Acronym: Preserve-HR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, Julio Nuñez, Principal Investigator, Clinical Professor, Fundación para la Investigación del Hospital Clínico de Valencia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BBLOQ-2017; 2017-005077-39 (EudraCT Number)
Record Dates: First submitted 2019-03-03; First posted 2019-03-12 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2020-07

CONDITIONS: Heart Failure With Normal Ejection Fraction; Chronotropic Incompetence
Keywords: Heart failure with preserved ejection fraction; Chronotropic incompetence; Functional capacity; Quality of life
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: This is a prospective, crossover, randomized (1:1) and single center study. After randomization, clinical and cardiac rhythm will be continuously registered during 30 days. The primary endpoint (peakVO2) will be assessed by CPET at 15 and 30-day in both groups. Patients with HFpEF, functional class NYHA II-III, chronic treatment with betablockers, and chronotropic incompetence will be enrolled. A sample size estimation [alfa: 0.05, power: 90%, a 15% loss rate, and delta change of mean peakVO2: +1.2 mL/kg/min (SD±2.5)] of 52 patients would be necessary to test our hypothesis.
Who Masked: Investigator
Masking Description: The examination tests will be performed by two blinded cardiologist to patients' allocation group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Active Comparator): Controlled Withdrawal of Beta-blockers and Cardiopulmonary Exercise Testing (CPET) Patient will be assessed for chronotr0pic incompetence by CPET. If the patient exhibits chronotropic incompetence, we will reduce half dose of previous beta-blocker.
  A cardiologist will evaluate clinically the the patient and the heart rate in 3 days. If clinical and heart rate stability (below 90 bpm), the patients will withdraw the beta-blocker and will be assessed by CPET at 15-day.
  After second CPET, the patient will introduce the half-dose of beta-blocker and will be evaluated in 3 days. If clinical stability, the patient will introduce the previous dose of beta-blocker A third CPET will be performed at 15-day
  Interventions: Drug: Controlled withdrawal of beta-blockers; Diagnostic Test: Cardiopulmonary Exercise Testing
- Arm B (Active Comparator): Cardiopulmonary Exercise Testing (CPET) and Controlled Withdrawal of Beta-blockers Patient will be assessed for chronotropic incompetence by CPET.If the patient exhibits chronotropic incompetence, a cardiologist will evaluate clinically the patient and the heart rate in 3 days and will be assessed by CPET at 15-day.
  After second CPET, the patient will reduce half dose of previous beta-blocker. A cardiologist will evaluate clinically the the patient and the heart rate in 3 days. If clinical and heart rate stability (below 90 bpm), the patients will withdraw the beta-blocker and will be assessed by CPET at 15-day.
  Interventions: Drug: Controlled withdrawal of beta-blockers; Diagnostic Test: Cardiopulmonary Exercise Testing

INTERVENTIONS:
Drug: Controlled withdrawal of beta-blockers — Controlled withdrawal of previos doses of beta-blockers after diagnosis of chronotropic incompetence
Diagnostic Test: Cardiopulmonary Exercise Testing — Cardiopulmonary Exercise Testing to evaluate the chronotropic incompetence and the primary endpoint (functional capacity)

SUMMARY:
The pathophysiology of heart failure with preserved ejection fraction (HFpEF) is complex and multifactorial. Chronotropic incompetence has emerged as a crucial mechanism, particularly in elderly patients. Betablockers, drugs with negative chronotropic effect, are commonly used in HFpEF, despite current evidence does not support its routine use in these patients. The aim of this work is to evaluate the effect of betablockers withdrawal in patients with HFpEF and chronotropic incompetence on functional capacity assessed by the peak oxygen consumption at maximal exercise (peakVO2) at 15 and 30 days after the intervention

DETAILED DESCRIPTION:
This is a prospective, crossover, randomized (1:1) and single center study. After randomization, clinical and cardiac rhythm will be continuously registered during 30 days. The primary endpoint (peakVO2) will be assessed by cardiopulmonary exercise testing (CPET) at 15 and 30-day in both groups. Patients with HFpEF, functional class NYHA II-III, chronic treatment with betablockers, and chronotropic incompetence will be enrolled. A sample size estimation [alfa: 0.05, power: 90%, a 15% loss rate, and delta change of mean peakVO2: +1.2 mL/kg/min (SD±2.5)] of 52 patients would be necessary to test our hypothesis.

In conclusion, optimizing therapy that improve quality of life and autonomy has become a health care priority in HFpEF. The investigators believe this study will add important knowledge for the treatment of a subgroup of HFpEF.

ELIGIBILITY:
Inclusion Criteria:

* Stable symptomatic patients with heart failure and preserved ejection fraction (NYHA class II-III).
* NT-proBNP >125 pg/mL in the last month
* Previous treatment with beta-blockers during the last 3 months
* Documented chronotropic incompetence, defined as: [(heart rate at peak exercise- heart rate at baseline)] / [(220 - age) - (heart rate at baseline)] < 0.62

Exclusion Criteria:

* Moderate to severe valvulopathy or miocardiopathy associated
* Patient with heart failure with recovered ejection fraction
* Acute Coronary Syndrome in the previous 12 months
* Angina or signs of myocardial ischemia on cardiopulmonary exercise testing
* Baseline heart rate>75 bpm.
* Uncontrolled hypertension, defined as >140mmHg systolic blood pressure and/or >90 mmHg diastolic blood pressure.
* Moderate to severe pulmonary disease associated
* Extracardiac comorbidity with a life expentancy less than 1 year.
* Unable to perform an adequate cardiopulmonary exersice test
* Previous treatment with digitalis or calcium channel blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2021-02-27 (Actual)

PRIMARY OUTCOMES:
Maximal functional capacity | The change in peak oxygen consumption will be measured at baseline, at 15-day and at 30-day
  Maximal functional capacity measured by peak oxygen consumption in the cardiopulmonary exercise testing (CPET). The peak oxygen consumption is expressed in mL/kg/min.The investigators will measure the change of peak oxygen consumption .

SECONDARY OUTCOMES:
Cognitive evaluation | The change in MMSE score will be measured at baseline, at 15-day and at 30-day
  We will asses the cognitive function by Mini Mental State Examination (MMSE) The MMSE is a cognitive test. The score is ranged from 0-30 (units of a scale). 30 points is the better outcome. The investigators will assess the change in the score.
Cognitive evaluation | The change in MoCa score will be measured at baseline, at 15-day and at 30-day
  We will asses the cognitive function by Montreal Cognitive Assessment (MoCa) The MoCa is a cognitive test. The score is ranged from 0-30 (units of a scale). 30 points is the better outcome. The investigators will assess the change in the score.
Quality of life evaluation | The change in MLHFQ score will be measured at baseline, at 15-day and at 30-day
  We will asses the quality of life by Minnesota living with heart failure questionnaire (MLHFQ). The MLHFQ is a quality of life questionnarie .The investigators will asses the changes in the full questionnarie. We will report the total score. The score is ranged from 0-105. 105 points is the worse outcome
Security: reporting on potential clinical adverse outcomes | Differences in the composite of adverse events between both arms will be measured at 15-day , at 30-day and 180-day
  Evaluation of adverse clinical outcomes during the study. The investigators will evaluate the composite of the following adverse events: mortality and/or readmissions due to cardiovascular reasons. The investigators will assess differences between both groups/arms

CONTACTS AND LOCATIONS:
Overall Officials: Julio Núñez, MD, PhD, Principal Investigator — Instituto de Investigacion Sanitaria INCLIVA
Locations (1):
- INCLIVA, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dominguez E, Palau P, Nunez E, Ramon JM, Lopez L, Melero J, Bellver A, Santas E, Chorro FJ, Nunez J. Heart rate response and functional capacity in patients with chronic heart failure with preserved ejection fraction. ESC Heart Fail. 2018 Aug;5(4):579-585. doi: 10.1002/ehf2.12281. Epub 2018 Mar 24. PMID 29573575
- [Background] Palau P, Dominguez E, Sanchis J, Bayes-Genis A, Nunez J. Heart Rate in Heart Failure With Preserved Ejection Fraction: Another Example of the Heterogeneity of This Syndrome. JACC Heart Fail. 2018 Apr;6(4):350-351. doi: 10.1016/j.jchf.2017.12.003. No abstract available. PMID 29598943
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Derived] Palau P, de la Espriella R, Seller J, Santas E, Dominguez E, Bodi V, Sanchis J, Nunez E, Bayes-Genis A, Bertomeu-Gonzalez V, Meyer M, Nunez J. beta-Blocker Withdrawal and Functional Capacity Improvement in Patients With Heart Failure With Preserved Ejection Fraction. JAMA Cardiol. 2024 Apr 1;9(4):392-396. doi: 10.1001/jamacardio.2023.5500. PMID 38324280
- [Derived] Palau P, Seller J, Dominguez E, Sastre C, Ramon JM, de La Espriella R, Santas E, Minana G, Bodi V, Sanchis J, Valle A, Chorro FJ, Llacer P, Bayes-Genis A, Nunez J. Effect of beta-Blocker Withdrawal on Functional Capacity in Heart Failure and Preserved Ejection Fraction. J Am Coll Cardiol. 2021 Nov 23;78(21):2042-2056. doi: 10.1016/j.jacc.2021.08.073. PMID 34794685
- [Derived] Palau P, Seller J, Dominguez E, Gomez I, Ramon JM, Sastre C, de la Espriella R, Santas E, Minana G, Chorro FJ, Gonzalez-Juanatey JR, Nunez J. Beta-blockers withdrawal in patients with heart failure with preserved ejection fraction and chronotropic incompetence: Effect on functional capacity rationale and study design of a prospective, randomized, controlled trial (The Preserve-HR trial). Clin Cardiol. 2020 May;43(5):423-429. doi: 10.1002/clc.23345. Epub 2020 Feb 19. PMID 32073676